CLINICAL TRIAL: NCT05483920
Title: Effects of Sleep Hygiene Education on Sleep Health in Community-Dwelling Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Black Hills State University (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Ashley Pfeiffer, Principal Investigator, Black Hills State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BlackHillsST; P20GM103443 (NIH)
Record Dates: First submitted 2022-07-29; First posted 2022-08-02 (Actual); Results first posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-02

CONDITIONS: Sleep Habit, Good; Sleep Hygiene; Health Behavior
MeSH Terms: conditions — Sleep Hygiene; Health Behavior

STUDY DESIGN:
Intervention Model Description: There will be two arms of the study including intervention and a control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One-time educational video (Experimental): A one-time educational video on best practices for good sleep hygiene
  Interventions: Behavioral: One-time educational video
- One-time educational video plus automated text messaging (Experimental): A one-time educational video on best practices for sleep hygiene plus daily automated text messages to reinforce habit.
  Interventions: Behavioral: One-time educational video plus automated text messaging

INTERVENTIONS:
Behavioral: One-time educational video — One-time educational video
  Arms: One-time educational video
Behavioral: One-time educational video plus automated text messaging — Educational video plus automated text messaging
  Arms: One-time educational video plus automated text messaging

SUMMARY:
This will be a study looking at trying to change community-dwelling older adults' behavior in regard to good sleep hygiene practices. Investigators will assess the efficacy through subjective outcome measures and objective physiological markers of good sleep through data collected with wearable technology devices.

DETAILED DESCRIPTION:
Community-dwelling older adults will be recruited and placed into one of two groups. Group one will watch a one-time educational video on sleep hygiene and group two will watch the video plus be sent daily automated text messages to reinforce the education learned in the video. The participants will receive the text messages for a total of 4 weeks. The control group will not receive any intervention during this time frame. Following the initial meeting, all participants will wear the sleep tracker on their wrists during the day and night for 4 weeks. The sleep tracker will monitor the physiological markers of sleep provided by wearable technology on sleep efficiency, time in bed, time actually sleeping, and time spent at each stage of sleep. At the end of the 4-week study period, the researchers will once again meet with each participant. The participant will complete the following questionnaires once again.

ELIGIBILITY:
Inclusion Criteria:

* Any adult between the ages of 50 and 80 will be recruited for the study

Exclusion Criteria:

* Anyone with a diagnosed sleep disorder such as insomnia or obstructive sleep apnea, and the inability to wear any sleep tracking device on their wrist.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashley M Pfeiffer, Principal Investigator — Black Hills State University
Locations (1):
- Black Hills State University, Spearfish, South Dakota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | One-time Educational Video | One-time Educational Video Plus Automated Text Messaging
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | One-time Educational Video | One-time Educational Video Plus Automated Text Messaging | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 7 | 11
  >=65 years | 11 | 8 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 14 | 27
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 14 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30
Sleep Hygiene Index [Mean (Full Range); unit: units on a scale] — sleep quality measurement. Scores range 0-21 with higher scores indicating poorer sleep quality. Collected through an electronic survey.
  units on a scale | 6.7 [2 to 15] | 8.7 [4 to 16] | 7.7 [2 to 16]

OUTCOME MEASURES:

1. Primary Outcome: Change Score From Baseline to 4-week Follow up on the Pittsburgh Sleep Quality Index
Description: Outcome measure for quality of sleep. Score ranges 0-21 with higher score equaling poor sleep quality
Time Frame: Baseline and 4-week follow up
Population: Change score average
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | One-time Educational Video | One-time Educational Video Plus Automated Text Messaging
Number analyzed (Participants) | 15 | 15
units on a scale | 1.6 [-1 to 7] | 2.5 [-1 to 10]

2. Primary Outcome: Change Score From Baseline to 4-week Follow up on the Sleep Hygiene Index
Description: Outcome measure for good sleep hygiene. Scores range from 0-52. Higher scores equate to worse sleep hygiene.
Time Frame: Baseline and 4-week follow up
Population: Average change scores
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | One-time Educational Video | One-time Educational Video Plus Automated Text Messaging
Number analyzed (Participants) | 15 | 15
units on a scale | 5.5 [-3 to 16] | 3.5 [-3 to 11]

3. Primary Outcome: Change Score From Baseline to 4-week Follow up on the Numeric Pain Rating Scale
Description: Outcome measure for average pain levels. Scores range from 0-10. Higher scores equate to higher pain levels.
Time Frame: Baseline and 4-week follow up
Population: Average change score
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | One-time Educational Video | One-time Educational Video Plus Automated Text Messaging
Number analyzed (Participants) | 15 | 15
units on a scale | 0.1 [-1 to 1] | 0.1 [-1 to 1]

4. Primary Outcome: Change Score From Baseline to 4-week Follow up on the Epworth Sleepiness Scale
Description: Outcome measure for average daytime sleepiness. Scores range from 0-24. Higher scores equate to worse daytime sleepiness.
Time Frame: Baseline and 4-week follow up
Population: average change score on ESS
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | One-time Educational Video | One-time Educational Video Plus Automated Text Messaging
Number analyzed (Participants) | 15 | 15
units on a scale | 1.3 [-4 to 8] | 2.3 [-1 to 8]

5. Primary Outcome: Change Score From Baseline to 4-weeks for Participants' Sleep Efficiency Using Wearable Technology.
Description: Sleep efficiency scores will be calculated using a sleep tracker device and are defined as time spent in bed versus time spent actually sleeping. 85% or higher is considered normal sleep efficiency. The average sleep efficiency score for the first three days at baseline and average sleep efficiency from the last 3 days of the 4 week study period will be used to gather the change score.
Time Frame: Baseline, 4-week follow up
Measure: Mean (Full Range); unit: percentage points of efficiency
Arm/Group | One-time Educational Video | One-time Educational Video Plus Automated Text Messaging
Number analyzed (Participants) | 15 | 15
percentage points of efficiency | -1.34 [-8.5 to 2.5] | -0.2 [-1.5 to 4]

6. Secondary Outcome: Change Score From Baseline to 4-week Follow up on the Perceived Stress Scale
Description: Outcome measure for average stress levels. Scores range from 0-40. The higher the score the worse the stress levels.
Time Frame: Baseline and 4-week follow up
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | One-time Educational Video | One-time Educational Video Plus Automated Text Messaging
Number analyzed (Participants) | 15 | 15
units on a scale | 3.1 [-2 to 13] | 1.9 [-10 to 9]

7. Secondary Outcome: Change Score From Baseline to 4-week Follow up on the Patient Specific Functional Scale
Description: Outcome measure for overall function. The participant chooses three functional day-to-day activities that they regularly participate in and they rate those activities from 0-10 on ease or difficulty of completing. 0 indicates unable to perform the activity, and 10 indicates no problem with the activity. The total score is calculated by adding all three activity scores and dividing by the number of activities listed for a total score ranging from 0-10.
Time Frame: Baseline and 4-week follow up
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | One-time Educational Video | One-time Educational Video Plus Automated Text Messaging
Number analyzed (Participants) | 15 | 15
units on a scale | 1.3 [-1.67 to 4.67] | 0.16 [-4.66 to 3.67]

8. Secondary Outcome: Change Scores From Baseline to 4-week Follow up for Participant's Body Mass Index
Description: Body mass index is measured by body weight [kg]/ height [m]2) from weight and height measurements to determine healthy body anthropometrics. Normal value is 18.5 to 24.9. Above these values is considered overweight and obese, under this is considered underweight.
Time Frame: baseline and 4-week follow up
Measure: Mean (Full Range); unit: kg/m^2 (kilograms/meters squared)
Arm/Group | One-time Educational Video | One-time Educational Video Plus Automated Text Messaging
Number analyzed (Participants) | 15 | 15
kg/m^2 (kilograms/meters squared) | -0.001 [-1.4 to 1.5] | 0.13 [-1.4 to 1.1]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored for the one-month of the study however no adverse events were reported.
Description: The number of participants at risk for serious adverse events, all-cause mortality, and other is zero due to a minimal risk activity of filling out surveys and wearing a sleep tracker.
Arm/Group | One-time Educational Video | One-time Educational Video Plus Automated Text Messaging
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

LIMITATIONS AND CAVEATS:
Limitations of the study include a small sample size, and minimal heterogeneity of gender, and race. We were limited to one geographical region.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-01): https://cdn.clinicaltrials.gov/large-docs/20/NCT05483920/Prot_SAP_000.pdf